CLINICAL TRIAL: NCT00328458
Title: A Phase I, Open-label, Dose-escalation, Safety Study of the Combination of EPO906 and Radiation Therapy for the Treatment of Patients With Cancer
Brief Title: EPO906 Plus Radiation Therapy for the Treatment of Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03C.275; 2003-33 (Other: CCRRC); JT 1035 (Other: JeffTrial Number)
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Central Nervous System Neoplasms; Head and Neck Neoplasms
Keywords: CNS and head and neck cancers; Histologically confirmed CNS malignancy head and neck; there is on standard therapy or; have failed standard therapy
MeSH Terms: conditions — Central Nervous System Neoplasms; Head and Neck Neoplasms | interventions — epothilone B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 Brain Tumors (Experimental): The investigational drug - EPO906 will be administered as an intravenous infusion over five to ten minutes on weeks 1, 3 and 6, for the duration of radiation therapy up to a maximum of 7 weeks. Duration of therapy will be determined by disease cohort.
  Interventions: Drug: EPO906 (epothilone B)
- Cohort 2 Head and Neck Tumors (Experimental): The investigational drug - EPO906 will be administered as an intravenous infusion over five to ten minutes on weeks 1, 3 and 6, for the duration of radiation therapy up to a maximum of 7 weeks. Duration of therapy will be determined by disease cohort.
  Interventions: Drug: EPO906 (epothilone B)

INTERVENTIONS:
Drug: EPO906 (epothilone B)

SUMMARY:
The purpose of this study is to determine the safety of the drug EPO906 that could shrink tumors when used with radiation therapy in cancer patients.

DETAILED DESCRIPTION:
* To determine the maximum tolerated dose (MTD) of EPO906 administered in combination with radiation therapy and establish a recommend phase II dose.
* To evaluate the safety and toxicity profile of EPO906 when administered concurrently with radiotherapy in three disease cohorts.
* To evaluate tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Requires a minimum of 3 weeks of radiation therapy
* Solid tumors with advanced or recurrent disease for which there is no standard therapy or tumors have failed standard therapy
* World Health Organization (WHO) performance status equal to or less than 2
* Life expectancy equal to or greater than 3 months

Exclusion Criteria:

* Any peripheral neuropathy
* Unresolved diarrhea greater than grade 1
* Patients who received any other investigational compound within the past 28 days
* Severe cardiac insufficiency
* Patients on Coumadin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-02; Primary Completion 2008-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of EPO906 | Baseline to 7 weeks

SECONDARY OUTCOMES:
Number of participants that successful complete 7 weekly cycles of EPO906 concurrently with radiotherapy | Baseline to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dicker, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org